CLINICAL TRIAL: NCT01709162
Title: A Randomized, Open-Label, Multicenter Phase II Study of Ipilimumab Retreatment Versus Chemotherapy for Subjects With Advanced Melanoma Who Progressed After Initially Achieving Disease Control With Ipilimumab Therapy
Brief Title: Study to Compare the Effect of Ipilimumab Retreatment With That of Chemotherapy in Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinued early due to enrollment challenges and changes in treatment standards
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-243; 2012-003291-38 (EudraCT Number)
Record Dates: First submitted 2012-10-12; First posted 2012-10-18 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ipilimumab, 3 mg/kg (Experimental): Participants received ipilimumab, 3 mg/kg, by intravenous infusion, every 3 weeks for a total of 4 doses or until disease progression, unacceptable toxicity, or withdrawal of consent
  Interventions: Biological: Ipilimumab
- Chemotherapy (Active Comparator): Participants received the investigator's choice of chemotherapy, administered per package instructions.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Biological: Ipilimumab
  Other Names: Yervoy; BMS-734016
  Arms: Ipilimumab, 3 mg/kg
Drug: Chemotherapy
  Arms: Chemotherapy

SUMMARY:
The purpose of the study is to determine whether additional doses of ipilimumab have a positive effect on survival in the treatment of advanced melanoma that has progressed after successful initial treatment with ipilimumab.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Key Inclusion Criteria:

* Histologic diagnosis of unresectable stage III or IV metastatic melanoma
* Prior ipilimumab induction treatment (3 mg/kg)
* Documented disease control [Stable Disease ≥3 months or Partial Response/Complete Response] after ipilimumab induction
* Documented progressive disease following disease control

Key Exclusion Criteria:

* Patients with brain metastasis are excluded, unless they are free of neurologic symptoms related to metastatic brain lesions and do not receive systemic corticosteroid therapy for the purpose of reducing intracranial inflammation in the 10 days prior to beginning retreatment with ipilimumab
* Any intervening anticancer therapy between last dose of ipilimumab induction and ipilimumab retreatment on study
* Patients who experienced any grade 3 immune-related adverse event (irAE) (except for endocrinopathies where clinical symptoms were controlled with appropriate hormone replacement therapy) or any grade 4 toxicity during prior treatment with ipilimumab
* Patients with a prior irAE that has not improved to grade 1 or better at randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (7):
  - Birmingham Hematology & Oncology Associates Llc, Birmingham, Alabama
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Investigative Clinical Research Of Indiana, Llc, Indianapolis, Indiana
  - Cancer Center Of Kansas, Wichita, Kansas
  - Comprehensive Cancer Center Of Nevada, Las Vegas, Nevada
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
- Local Institution, Vienna, Austria
- France (3):
  - Local Institution, Bordeaux
  - Local Institution, Nantes
  - Local Institution, Paris
- Germany (5):
  - Local Institution, Cologne
  - Local Institution, Erfurt
  - Local Institution, Göttingen
  - Local Institution, Heidelberg
  - Local Institution, Kiel
- Local Institution, Siena, Italy

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 31 participants were enrolled. Of the 23 who were randomized, 22 received treatment .
Groups:
- Ipilimumab, 3 mg/kg: Participants received ipilimumab, 3 mg/kg, intravenously by infusion every 3 weeks for a total of 4 doses or until disease progression, unacceptable toxicity, or withdrawal of consent
- Chemotherapy: Participants received the investigator's choice of chemotherapy, dosed per package instructions.
Period: Overall Study
Arm/Group | Ipilimumab, 3 mg/kg | Chemotherapy
Started | 18 (Randomized) | 5 (Randomized)
Received Treatment | 18 | 4
Still Receiving Treatment | 0 | 0
Completed | 12 (Completed treatment as per protocol) | 0 (Completed treatment as per protocol)
Not Completed | 6 | 5
Not completed — Disease progression | 3 | 3
Not completed — Study drug toxicity | 2 | 0
Not completed — Administrative reason by sponsor | 0 | 1
Not completed — Other | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab, 3 mg/kg | Chemotherapy | Total
Number analyzed (Participants) | 18 | 5 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (11.38) | 64.2 (4.32) | 62.7 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 12 | 4 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 18 | 5 | 23
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — ECOG is a 6-item scale used to assess disease progression, daily functioning, appropriate treatment, and prognosis. Performance status is scored on a scale ranging from 0-5, with (best score) 0=fully active and able to carry on all predisease performance without restriction and (worst score) 5=death.
  Participants
    0 | 13 | 5 | 18
    1 | 5 | 0 | 5
Disease Stage at Study Entry [Number; unit: Participants] — By the American Joint Committee on Cancer staging: Stage 1=no spread to lymph nodes/organs, <1 mm thick and not ulcerated (1A) or <1 mm thick and ulcerated or 1-2 mm thick and not ulcerated (1B). Stage 2=no spread to lymph nodes (LN) or other organs, 1-2 mm thick and ulcerated or 2-4 mm thick and not ulcerated (2A) or 2-4 mm thick and ulcerated or >4 mm thick and not ulcerated (2B), or >4 mm thick and ulcerated (2C). Stage 3 (A,B,C)=any thickness, ulcerated or not, and spread to nearby LN or nearby tissue but not LN. Stage 4=spread to LN, other organs, or areas far from original tumor site.
  Participants
    Stage III | 1 | 1 | 2
    Stage IV | 17 | 4 | 21
Objective Response to Prior Ipilimumab Treatment [Number; unit: Participants] — Tumors assessed per Response Evaluation Criteria In Solid Tumors Criteria for target lesions: Complete response (CR)=disappearance of all target lesions. Partial response (PR)=30% or greater decrease in sum of the longest diameter (LD) of target lesions. Progressive disease (PD)=a 20% or greater increase in sum of the LD of all target lesions, taking as reference the smallest sum LD recorded at or following baseline. Stable disease=neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. Objective response=number of patients with best response of CR or PR.
  Participants
    Complete response/Partial response | 6 | 0 | 6
    Stable disease | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined for each patient as the time between randomization and death. If a patient has not died, he or she will be censored at the time of last contact (last known alive date)
Time Frame: From randomization to death or last known alive date, assessed up to 15.6 months
Population: All participants who were randomized
Measure: Median (Full Range); unit: Months
Arm/Group | Ipilimumab, 3 mg/kg | Chemotherapy
Number analyzed (Participants) | 18 | 5
Months | 6.3 [3.2 to 15.6] | 3.1 [0.0 to 8.6]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined per arm as the total number of randomized participants with best overall response as complete response, partial response, or stable disease, divided by the total number of randomized participants in the arm. Bristol-Myers Squibb terminated this study early because the study would not meet its scientific objective in the predefined time frame. Thus, no participants were analyzed. Because the study ended before best overall response could be determined, no participants were analyzed.
Time Frame: Every 3 months for approximately 3.5 years after start of randomization and then every 6 months until confirmed and documented progressive disease
Population: All participants who were randomized
Arm/Group | Ipilimumab, 3 mg/kg | Chemotherapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Best Overall Response Rate (BORR)
Description: BORR is defined per arm as the total number of randomized patients with a best overall response of complete response or partial response, divided by the total number of randomized patients in the arm. Bristol-Myers Squibb terminated this study early because the study would not meet its scientific objective in the predefined timeframe. Because the study ended before best overall response for all patients was defined, no participant data was analyzed.
Time Frame: as for outcome 2
Population: All participants who were randomized
Arm/Group | Ipilimumab, 3 mg/kg | Chemotherapy
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, and Immune-related AEs (irAEs)
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: From Day 1 of treatment to 90 days after last dose (or to death date for death information)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ipilimumab, 3 mg/kg | Chemotherapy
Number analyzed (Participants) | 18 | 4
Participants
  Deaths | 5 | 1
  Deaths within 90 days of last dose | 1 | 0
  AEs leading to discontinuation | 2 | 0
  SAEs | 7 | 0
  irAEs | 10 | 1

ADVERSE EVENTS:
Groups:
- Ipilimumab, 3 mg/kg: Participants received ipilimumab, 3 mg/kg, by intravenous infusion every 3 weeks for a total of 4 doses or until disease progression, unacceptable toxicity, or withdrawal of consent
Arm/Group | Ipilimumab, 3 mg/kg | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 7/18 | 0/4
Other Adverse Events (participants affected / at risk) | 15/18 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab, 3 mg/kg (N=18) | Chemotherapy (N=4)
Depression (Psychiatric disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab, 3 mg/kg (N=18) | Chemotherapy (N=4)
Hypotension (Vascular disorders) | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Otitis media (Infections and infestations) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood corticotrophin decreased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Asthenia (General disorders) | 3 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Oedema peripheral (General disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Fatigue (General disorders) | 4 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
As planned, accrual of participants was to be completed within 21 months. However, current projections showed that 4 to 5 years were needed. The study was terminated early because the scientific objective could not be met in the predefined timeframe.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.